CLINICAL TRIAL: NCT03486158
Title: Optimalization of Disease Control and Quality of Life in Inflammatory Bowel Disease Using e-Health Measurements Via a Smart Phone Application; CalproSmart
Brief Title: The CalproSmartNOR Study - a New Clinical Tool for Monitoring Patients With Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Møre og Romsdal HF (Other Government)
Collaborators: Alesund Hospital (Other); Calpro AS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017/1792
Record Dates: First submitted 2018-03-27; First posted 2018-04-03 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Leukocyte L1 Antigen Complex; Feces; Cell Phone; Biomarkers; Recurrence; Prognosis; Clinical Chemistry Tests
MeSH Terms: conditions — Inflammatory Bowel Diseases; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CalproSmart application (Experimental): In addition to regular outpatient clinic visits and a routine CalproSmart test every 3 months, patients are instructed to obtain fecal samples if they experience symptoms suspect of recurrent IBD and to perform home analysis with CalproSmart™ system test kit
  Interventions: Device: CalproSmart™ system
- Standard follow-up (No Intervention): In addition to regular outpatient clinic visits and a routine calprotectin test in the same week as the visit date, patients bring home an Fecal-calprotectin tube and envelope and are instructed to obtain fecal samples and send these to local lab if they experience symptoms suspect of recurrent IBD

INTERVENTIONS:
Device: CalproSmart™ system — Home test kit for measurement of calprotectin in fecal samples. A new clinical tool for monitoring patients with inflammatory bowel disease, enabling measurement of calprotectin level of rapid test through a specially developed Smartphone application (platforms such as Android o Iphone)
  Arms: CalproSmart application

SUMMARY:
The aim of this study is to prove that getting immediate calprotectin test results on the patients Smartphone (platforms such as Android or Iphone), will both stimulate patients with inflammatory bowel disease (IBD) to closer follow up of their disease, and that immediate automatic e-mails to a IBD-nurse will lead to earlier decision-making on further treatment and follow-up by health personnel (optimized medication, endoscopy etc).

DETAILED DESCRIPTION:
There has been a shift in the therapeutic approach for inflammatory bowel disease (IBD) from symptom-tailored towards inflammation-targeted treatments. Mucosal healing, although not well-defined in past literature, is an objective marker of improvement as well as of favorable prognosis, not only in trials but also in routine clinical practice. However, utilization of frequent endoscopic procedures to assess mucosal healing would be a burden to patients and the stretched endoscopic services in the national health services. A non-invasive marker would give the opportunity to patients and physicians to titrate treatment to inflammatory activity with the aspiration to change the course of the disease.

Calprotectin (FCALP) is a calcium-binding protein abundant in the cytoplasm of neutrophils and macrophages that can be measured in feces reliably. Samples can be transported or stored at room temperature for at least 3 days. FCALP correlates well with histological and endoscopic disease activity in ulcerative colitis and radiology in Crohn's disease.

More importantly calprotectin predicts clinical relapse, outperforming other common non-invasive markers of inflammation (CRP, ESR), and it may also outperform endoscopy in predicting short and long term relapse.

Patients are currently required to provide a stool sample in a universal (non-specialized) container, which usually is processed in a central laboratory. The container is a small plastic cylinder secured with a screw top which has a longitudinal scoop attached to its inner surface. In order to collect the sample, the patients usually put some toilet paper in the toilet and after defecating use the scoop to collect the fecal sample. Then the container is brought to hospital in person and is processed by the laboratory staff. This is a laborious process, as a certain quantity of fecal material has to be manually extracted from each individual sample using a separate kit prior to the measurement, which is performed using an ELISA kit.

In relation to e-Health telemedicine's increasing importance as an aid to therapeutic approaches for IBD patients, the need for an accurate and user-friendly home test for measuring fecal calprotectin concentration has emerged. New technology has improved the collection device, and simplified the collection process by providing a paper sampler device placed over the toilet bowel, making the sampling both easier and cleaner. A preferred system should easily been able to convert the sample into an extract, measure the calprotectin concentration with a rapid-test read by a smartphone application (platforms such as Android or Iphone), to produce an instant result for the patient at home which also concomitantly and securely should be sent via a portal to the treating clinician.

The CalproSmart™ system is a Home test kit for measurement of calprotectin in fecal samples, and a new clinical tool for monitoring patients with inflammatory bowel disease. The system consists of five components and a Smartphone - application (platforms such as Android or Iphone); A) A sampler and nitrile gloves for collecting stool samples B) A prefilled extraction device to collect stool sample C) A lateral-flow rapid test D) A support frame with a design that enables measurement of calprotectin level of rapid test through a specially developed Smartphone application (platforms such as Android or Iphone).

ELIGIBILITY:
Inclusion Criteria:

* Ulcerative colitis and Crohns disease diagnosis that fulfil the international Copenhagen diagnostic criteria for inflammatory bowel diseases (IBD)
* Remission, mild or moderate disease activity defined as 6-point Mayo Score <= 3 or Harvey Bradshaw index (HBI) <= 16
* Written and oral consent about participation in the project
* In a mental and physical state in which every step of the procedure is understood and feasible
* Ability to obtain and prepare a fecal sample and to use the Smartphone application (platforms such as Android or Iphone)

Exclusion Criteria:

* Severe disease activity defined as 6-point Mayo Score > 3 or HBI > 16
* Unable to read, understand or perform one or several steps of the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2020-03-27 (Actual)

PRIMARY OUTCOMES:
Change in disease activity index 1 | At baseline 3, 6, 9 and 12 months according to randomization arm
  Crohn disease and Ulcerative colitis acidity measured using the Harvey-Bradshaw index ( total score 0-20 points, where < than 3 indicate remission and > 7 indicates severe disease ) and 6 point Mayo Score (total score 0-6, > 2 indicates moderate to severe disease.
Change in disease activity index 2 | At baseline, 3, 6, 9 and 12 months according to randomization arm
  Fecal Calprotectin (mg/kg) where < 50 indicates no activity, 50-200 remission and > 250 activity - moderate to severe

SECONDARY OUTCOMES:
Time to disease flare | At 3, 6, 9 and 12 months according to randomization arm
  Patients in remission at baseline visit
Time to remission | At 3, 6, 9 and 12 months according to randomization arm
  Patients with mild to moderate disease activity in the course of the study
Quality of life according to disease activity | At baseline and at 12 months
  The Norwegian validation study (N-IBDQ) revealed a five-dimensional structure: emotional function-1 (fatigue, energy), bowel function-1 (stool consistency and pattern), bowel function-2 (bowel pain and discomfort), social function (work attendance, cancelling social events) and emotional function-2 (worries). All of the responses were scored on a 7-point Likert Scale, with a score of 7 representing no problems and a score of 1 representing severe problems. This gives a possible score range of 32-224, with a higher score reflecting improved HRQoL
Hospitalization | At 3, 6, 9 and 12 months
  Number of admission to hospital care due to disease activity
Outpatient clinic contacts | At 3, 6, 9 and 12 months
  Number of contacts to the outpatient clinic care due to disease activity
Work activity | At 3, 6, 9 and 12 months
  Assessed by number of presenteeism /absenteeism at work

CONTACTS AND LOCATIONS:
Overall Officials: Dag Arne Lihaug Hoff, md phd, Study Director — Helse Møre & Romsdal HF, Ålesund Hospital
Locations (1):
- The Outpatient Clinic, Department of gastroenterology, Ålesund Hospital, Helse Møre og Romsdal HF, Ålesund, Norway

IPD SHARING:
Plan to Share IPD: No